CLINICAL TRIAL: NCT04764279
Title: Rural-specific OPTIFAST Intervention - A Randomized Study for Partial Remission of Type 2 Diabetes in Patients With Obesity Between the Age of 18 and 65
Brief Title: A Rural OPTIFAST Intervention for Partial Remission of Type 2 Diabetes in Adults With Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Marathon Family Health Team (Other)
Responsible Party: Principal Investigator, Dr. Megen Brunskill, Principal Investigator, Marathon Family Health Team
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-20-3
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Diabetes Mellitus, Type 2; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Intervention Model Description: A two arm, open-label randomized study will be conducted with a total of 30 patients being randomly assigned (1:1) to either of the two study arms: VLCD ( OPTIFAST®) intervention or best-practice care (control). The sample size was determined assuming a 46% partial remission rate of DMII in the VLCD group at year 1 and 4% in the usual care group and power of 80%. These rates are based on the findings of the DiRECT study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OPTIFAST Arm (Experimental): Participants in the intervention group will be given OPTIFAST® meal replacement shakes, 4 per day to achieve 900kcal/day, for the first 12 weeks of the study. The second phase will consist of partial meal replacement and food reintroduction over a 4 week period. When the intervention group begins to reintroduce foods, all study participants will be provided a workbook, created for the study, to explain optimal lifestyle changes for DMII management. The third phase will be a 8-month follow-up of participants on continued healthy lifestyle as described in the workbook.
  Interventions: Dietary Supplement: OPTIFAST dietary supplement
- Control/Usual Care Arm (No Intervention): Usual Care : A gift card will be offered to participants in the control group to stabilize the incentive of the intervention. Participants in the control group will receive usual diabetes care based on the current Canadian Diabetes Association guidelines by their family physician. Participants in the control group will receive the same workbook as the intervention group at 16 weeks into the study.

INTERVENTIONS:
Dietary Supplement: OPTIFAST dietary supplement — Participants will use Optifast Nutrition Supplement as previously described
  Arms: OPTIFAST Arm

SUMMARY:
As rural Canada is a resource poor health service environment, we propose to test whether an OPTIFAST dietary replacement intervention, without the service intensive behavioural component, can cause partial remission of DMII in patients with obesity and DMII.

DETAILED DESCRIPTION:
The objective of this study is to see if a rural-specific OPTIFAST intervention, of dietary replacement only, can cause a partial remission of DMII patients with obesity between the age of 18 and 65 diagnosed with DMII within the last 6 years. The goal is to inform the current diabetes routine care by standardizing a rural protocol on the effectiveness of rural-specific OPTIFAST intervention for people with DMII who want to attain partial remission of DMII.

ELIGIBILITY:
Inclusion Criteria:

* Study participants will be patients of the MFHT, aged 18 to 65, BMI between 27 and 45 kg/m 2 , and newly diagnosed with DMII within the past 6 years.

Exclusion Criteria:

* The exclusion criteria will be anti-hyperglycemic medications, slow onset of type 1 diabetes (DMI) or maturity onset diabetes of the young (MODY), renal dysfunction (serum creatinine>150 μmol/l), history of myocardial infarction, untreated thyroid disease, consumption of 4 alcohol units/day by men and 3 units/day by women, chronic steroid consumption, unstable psychiatric conditions, and atypical antipsychotic medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Partial Remission of Diabetes | 12 months
  HbA1c<6.5% without antihyperglycemic medications

SECONDARY OUTCOMES:
Improved Insulin Resistance | 12 months
  Reduction of Fasting Insulin
Improved Blood Pressure | 12 months
  Reduction in blood pressure measures
Weight loss | 12 months
  Reduction in BMI
Reduction in Visceral Adiposity | 12 months
  Reduction in waist circumference

CONTACTS AND LOCATIONS:
Overall Officials: Megen T Brunskill, MD, Principal Investigator — Marathon Family Health Team

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Athinarayanan SJ, Adams RN, Hallberg SJ, McKenzie AL, Bhanpuri NH, Campbell WW, Volek JS, Phinney SD, McCarter JP. Long-Term Effects of a Novel Continuous Remote Care Intervention Including Nutritional Ketosis for the Management of Type 2 Diabetes: A 2-Year Non-randomized Clinical Trial. Front Endocrinol (Lausanne). 2019 Jun 5;10:348. doi: 10.3389/fendo.2019.00348. eCollection 2019. PMID 31231311
- [Background] Ard JD, Lewis KH, Rothberg A, Auriemma A, Coburn SL, Cohen SS, Loper J, Matarese L, Pories WJ, Periman S. Effectiveness of a Total Meal Replacement Program (OPTIFAST Program) on Weight Loss: Results from the OPTIWIN Study. Obesity (Silver Spring). 2019 Jan;27(1):22-29. doi: 10.1002/oby.22303. Epub 2018 Nov 13. PMID 30421863
- [Background] Bilandzic A, Rosella L. The cost of diabetes in Canada over 10 years: applying attributable health care costs to a diabetes incidence prediction model. Health Promot Chronic Dis Prev Can. 2017 Feb;37(2):49-53. doi: 10.24095/hpcdp.37.2.03. PMID 28273040
- [Background] Leslie WS, Taylor R, Harris L, Lean ME. Weight losses with low-energy formula diets in obese patients with and without type 2 diabetes: systematic review and meta-analysis. Int J Obes (Lond). 2017 Jan;41(1):96-101. doi: 10.1038/ijo.2016.175. Epub 2015 Oct 4. PMID 27698345
- [Background] Pohar SL, Majumdar SR, Johnson JA. Health care costs and mortality for Canadian urban and rural patients with diabetes: population-based trends from 1993-2001. Clin Ther. 2007;29 Spec No:1316-24. PMID 18046931
- [Background] Supina AL, Guirguis LM, Majumdar SR, Lewanczuk RZ, Lee TK, Toth EL, Johnson JA. Treatment gaps for hypertension management in rural Canadian patients with type 2 diabetes mellitus. Clin Ther. 2004 Apr;26(4):598-606. doi: 10.1016/s0149-2918(04)90062-8. PMID 15189757
- [Background] Hallberg SJ, Gershuni VM, Hazbun TL, Athinarayanan SJ. Reversing Type 2 Diabetes: A Narrative Review of the Evidence. Nutrients. 2019 Apr 1;11(4):766. doi: 10.3390/nu11040766. PMID 30939855
- [Background] Lean ME, Leslie WS, Barnes AC, Brosnahan N, Thom G, McCombie L, Peters C, Zhyzhneuskaya S, Al-Mrabeh A, Hollingsworth KG, Rodrigues AM, Rehackova L, Adamson AJ, Sniehotta FF, Mathers JC, Ross HM, McIlvenna Y, Stefanetti R, Trenell M, Welsh P, Kean S, Ford I, McConnachie A, Sattar N, Taylor R. Primary care-led weight management for remission of type 2 diabetes (DiRECT): an open-label, cluster-randomised trial. Lancet. 2018 Feb 10;391(10120):541-551. doi: 10.1016/S0140-6736(17)33102-1. Epub 2017 Dec 5. PMID 29221645
- [Background] Lewis MC, Phillips ML, Slavotinek JP, Kow L, Thompson CH, Toouli J. Change in liver size and fat content after treatment with Optifast very low calorie diet. Obes Surg. 2006 Jun;16(6):697-701. doi: 10.1381/096089206777346682. PMID 16756727
- [Background] Miura J, Arai K, Tsukahara S, Ohno M, Ikeda Y. The long term effectiveness of combined therapy by behavior modification and very low calorie diet: 2 years follow-up. Int J Obes. 1989;13 Suppl 2:73-7. PMID 2613431
- [Background] Yawn BP, Casey M, Hebert P. The rural health care workforce implications of practice guideline implementation. Med Care. 1999 Mar;37(3):259-69. doi: 10.1097/00005650-199903000-00006. PMID 10098570
- [Background] O'Neil PM, Miller-Kovach K, Tuerk PW, Becker LE, Wadden TA, Fujioka K, Hollander PL, Kushner RF, Timothy Garvey W, Rubino DM, Malcolm RJ, Weiss D, Raum WJ, Salyer JL, Hermayer KL, Rost SL, Veliko JL, Sora ND. Randomized controlled trial of a nationally available weight control program tailored for adults with type 2 diabetes. Obesity (Silver Spring). 2016 Nov;24(11):2269-2277. doi: 10.1002/oby.21616. PMID 27804264
- See also: Canadian Diabetes Strategy — https://www.ourcommons.ca/Content/Committee/421/HESA/Reports/RP10365941/hesarp23/hesarp23-e.pdf
- See also: Reversibility of Type 2 Diabetes — https://search-proquest-com.proxy1.lib.uwo.ca/docview/1885883419?accountid=15115&pq-origsite=summon